CLINICAL TRIAL: NCT07092501
Title: An Experimental Evaluation of Menthol-Flavored Tobacco Accessories: Subjective Effects and Purchasing Behavior
Brief Title: An Experimental Evaluation of Menthol-Flavored Tobacco Accessories
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: VT IRB # 25-695
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2025-07

CONDITIONS: Cigarette; Smoking Behaviors; Cigarette Smoking Behavior
Keywords: Menthol Cigarettes; Subjective Ratings; Experimental Tobacco Marketplace; Menthol Accessories
MeSH Terms: conditions — Smoking; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Menthol cigarette smokers (Experimental): Menthol cigarette smokers will sample non-menthol cigarettes mentholated using menthol-flavored accessories (e.g., crush balls, filter tips, aroma cards), non-menthol cigarettes and their own cigarettes. Participants will provide subjective ratings of each product (e.g., liking, strength, ease of use) in comparison to their usual menthol cigarette brand. They will complete hypothetical cross-commodity purchase tasks and ETM trials to assess product demand and likelihood of use in different conditions.
  Interventions: Behavioral: Mentholated cigarette sampling; Behavioral: Hypothetical Policy Scenarios; Behavioral: Subjective value assessment

INTERVENTIONS:
Behavioral: Mentholated cigarette sampling — Participants will participate in five sampling trials (menthol cigarette, non-menthol cigarette, non-menthol cigarette mentholated with accessory 1, with accessory 2, and with accessory 3). They will be exposed to these trials in a randomized order. In each trial, participants will take four guided puffs from one cigarette. They will have a 20-minute washout period between trials. They will first complete subjective ratings for the product they just sampled. Then, during the washout period, participants will be instructed to rinse their mouth thoroughly with room-temperature water three times. Each rinse will last approximately 10 seconds, and participants will be guided to swish the water around all areas of the mouth before expectorating. A one-minute rest will follow each rinse to allow residual taste to dissipate. No food or drink will be allowed during this period.
Behavioral: Hypothetical Policy Scenarios — Participants will complete the real Experimental Tobacco Marketplace consisting of one control trial and two menthol flavor restrictions (menthol cigarettes unavailable and both menthol cigarettes and menthol-flavored accessories unavailable). Participants will complete a total of 3 purchasing trials each for 7 days worth of products. In each trial, participants will buy tobacco products to use throughout the next 7 days. At the end of the session, the participant will randomly draw an individual purchasing trial and will receive all the products purchased at that trial to use over the next week. During the following 7 days, the participant is asked to use only the tobacco/nicotine products received during the study.
Behavioral: Subjective value assessment — Participants will complete a hypothetical purchase task where the price of a variety of products will increase progressively during the task.

SUMMARY:
In a within-subjects design in-laboratory study, participants will sample non-menthol cigarettes mentholated with various accessories (e.g., crush balls, filter tips, aroma cards) in a controlled setting. They will compare these to their preferred menthol brand using subjective ratings (e.g., liking, strength, ease of use) and complete purchase tasks and ETM trials to assess product demand and likelihood of future use.

DETAILED DESCRIPTION:
Cigarette smoking remains the leading preventable cause of death and disease in the United States (US), accounting for half a million deaths per year and nearly 30% of all cancer deaths. More than 28 million US adults smoke daily, 35% of whom smoke menthol flavored cigarettes. Menthol cigarettes are linked to increased risk of smoking initiation and reduced likelihood of cessation. In addition to increased product appeal and attractiveness, menthol's cooling properties may induce misperceptions of reduced harm and mask early symptoms of respiratory disease. A cohort study (N ≈ 1 million) by the American Cancer Society found that former menthol smokers had a 12-43% higher risk of all-cause and heart disease mortality compared to former non-menthol smokers.

Efforts to reduce the appeal of cigarettes have been enacted worldwide, with several countries adopting regulatory policies on menthol flavor in tobacco products. In the US, state and local governments have been leading these tobacco control efforts, with over 140 localities implementing a menthol cigarette ban as of December 2024, including California and Massachusetts. Menthol bans have been effective in reducing smoking prevalence and increasing cessation rates. Nonetheless, at least one-third of menthol smokers continue to smoke after a menthol ban. A key contributor is the tobacco industry's promotion of mentholation accessories - including crush balls, filter tips, aroma cards - that consumers can use to flavor non-menthol cigarettes after purchase. These accessories, often nicotine-free and sold separately from tobacco products, fall outside the scope of tobacco regulations and have grown in popularity in jurisdictions with bans. Studies indicate that up to 40% of pre-ban menthol smokers may adopt these accessories after restrictions take effect, undermining public health objectives.

In this study, the investigators will experimentally examine subjective ratings of non-menthol cigarettes, flavored with various menthol-flavor accessories (e.g., crush balls, filter tips, aroma cards), compared to participants' own preferred brand of menthol cigarettes and non-menthol cigarettes equivalent.

In a within-subject design, menthol cigarette smokers will sample non-menthol cigarettes mentholated with menthol-flavor accessories (e.g., crush balls, filter tips, aroma cards), non-menthol cigarettes and their own cigarettes. Participants will provide subjective ratings of each product (e.g., liking, strength, ease of use) in comparison to their usual menthol cigarette brand. They will complete hypothetical cross-commodity purchase tasks and will complete one control trial and two ETM conditions representing different levels of restriction on menthol flavor in cigarettes. Within each condition, the investigators will manipulate availability of products and observe purchasing patterns across tobacco products and menthol-flavored accessories.

The study will consist of one in-lab visit. The study phases include: 1) Screening Phase; 2) Consent and assessments; 3) Sampling and subjective ratings assessments, and 4) ETM and hypothetical purchasing trials.

1. Screening phase Recruited participants will be redirected to an online pre-screening platform (e.g., Ripple) to complete assessments related to tobacco and nicotine use, pregnancy status (if applicable), physical and medical conditions, use of smoking cessation medications, intentions to quit tobacco or nicotine products, and plans to relocate from the area. Individuals who meet the eligibility criteria will be invited to participate in the full research study. Participants will also report on cigarette brand preferences for preparation of the research cigarettes to be sampled.

   1.1) Cigarette preparation: In this project, participants' preferred brand of cigarettes will be used for sampling. They will sample their preferred menthol cigarette, a non-menthol equivalent and the non-menthol equivalent flavored with two different types of menthol-flavored accessories. All external indicators of whether a cigarette is menthol or non-menthol will be carefully concealed to prevent participants from identifying the product type based on visual cues. Fisherbrand Labeling Tape (non-toxic, heat-resistent, 13mm wide; Fisher Scientific, Pittsburgh, PA) will be used to cover any identifying marks near the filter end, without obstructing the filter vent holes. If markings are present along the tobacco rod, they will be further masked using top-brand cigarette papers. This procedure ensures that participants are blind to the menthol status of the cigarette, maintaining the integrity of experimental conditions.
2. Consent and Assessments (approximately 1 hour) In the consent and initial assessment session, participants will go through standard consent procedures. Participants will provide a breath sample to confirm recent levels of smoking that will be measured using a CoVita® Micro+ Basic Smokerlyzer. Participants of childbearing potential will be asked to provide a urine sample for pregnancy testing. Those with a positive pregnancy result will be excluded from the study. Participants will complete a timeline follow back to assess the previous month's smoking habits and consumption of nicotine products to determine ETM budget. Participants will complete a survey with demographic questions and nicotine/tobacco-related assessments (Fagerstrom Test for Cigarette Dependence, Perceived Health Risk adapted, Questionnaire on Smoking Urges-Brief, Motivation to Quit, Self-efficacy to Quit, and The Contemplation Ladder adapted).
3. Sampling and subjective ratings assessments (approximately 2:30 hours) . Participants will participate in five sampling trials (menthol cigarette, non-menthol cigarette, non-menthol cigarette mentholated with accessory 1, with accessory 2, and with accessory 3). They will be exposed to these trials in a randomized order. In each trial, participants will take four guided puffs from one cigarette. They will have a 20-minute washout period between trials. They will first complete subjective ratings for the product they just sampled. Then, during the washout period, participants will be instructed to rinse their mouth thoroughly with room-temperature water three times. Each rinse will last approximately 10 seconds, and participants will be guided to swish the water around all areas of the mouth before expectorating. A one-minute rest will follow each rinse to allow residual taste to dissipate. No food or drink will be allowed during this period.
4. ETM and hypothetical purchasing trials (approximately 30 minutes).

In the ETM session, participants will be provided with an individual 7-day experimental budget calculated based on their average tobacco/nicotine consumption over the past 7 days. For example, if a participant reports smoking 20 cigarettes per day (a pack), they will receive $70.00, equivalent to 140 cigarettes (or 7 packs) multiplied by $0.50 per cigarette (market price of an individual cigarette) to spend in the ETM. In the ETM, first, participants will experience two practice trials. Then, participants will complete the real ETM consisting of one control trial and two menthol flavor restrictions (menthol cigarettes unavailable and both menthol cigarettes and menthol-flavored accessories unavailable). Participants will complete a total of 3 purchasing trials each for 7 days worth of products. In each trial, participants will buy tobacco products to use throughout the next 7 days. At the end of the session, the participant will randomly draw an individual purchasing trial and will receive all the products purchased at that trial to use over the next week. During the following 7 days, the participant is asked to use only the tobacco/nicotine products received during the study.

The investigators will use repeated-measures analysis of variance (ANOVA) to assess differences in subjective ratings (e.g., liking, strength, ease of use) and purchasing behavior across the five product types. Main effects and planned comparisons will be tested to determine whether menthol accessories significantly alter product perceptions or demand compared to non-menthol cigarettes and usual menthol brands.

Purchasing behavior from the ETM trials and hypothetical purchase tasks will be analyzed using generalized linear mixed models (GLMMs) to account for repeated observations within individuals and the categorical nature of product selections. Demand metrics (e.g., breakpoint, elasticity, intensity) will be derived from purchase task data using established demand curve modeling procedures.

Exploratory analyses will examine the moderating effects of demographic variables (e.g., age, gender, race/ethnicity) and baseline smoking behavior (e.g., cigarettes per day, brand preference) on product perceptions and purchasing patterns. All analyses will be conducted using R, with significance set at p < .05 and adjustments made for multiple comparisons where applicable.

Additional analysis may be conducted.

ELIGIBILITY:
Inclusion criteria:

* Provide informed consent
* Be a menthol cigarette smoker
* Be at least 21 years of age or older
* Provide a breath sample for measuring carbon monoxide (CO ≥ 8 ppm)
* Smoke at least 10 cigarettes daily
* Use other tobacco products less than weekly

Exclusion criteria:

* Have uncontrolled physical or mental health conditions
* Use of smoking cessation medications (e.g., nicotine replacement, bupropion, varenicline) in the past 30 days
* Report concrete, immediate plans to alter/quit using their usual tobacco products in the next 30 days
* If they are pregnant or lactating
* Have plans to move out of the area during the experiment

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Modified Cigarette Evaluation Questionnaire (mCEQ) | Day 1
  Participants will provide the subjective ratings (e.g. liking, strength, ease of use) of each product in comparison to their usual menthol cigarette brand. The scale ranges from not at all (1) to extremely (7). Four factor scoring comprising stimulant effects (sum of items 5, 7 and 8, range from 3 to 21), positive reinforcement (sum of items 2, 3 and 12, range from 3 to 21), negative reinforcement (sum of items 4, 6 and 11, range from 3 to 21) and aversion (sum of items 9 and 10, range from 2 to 14). High scores represents higher positive effects for the first 3 factor and higher negative effect for the last factor.

SECONDARY OUTCOMES:
Own-price and cross-price demand intensity (q0) | Day 1
  Participants will complete purchasing trials in a hypothetical purchase task. In the hypothetical purchase task, participants will complete multiple trials where the price of a product will increase progressively. The availability of alternative products will be manipulated. We will measure demand intensity (q0) while product prices increase across trials.
Own-price and cross-price demand elasticity (alpha) | Day 1
  Participants will complete purchasing trials in a hypothetical purchase task. In the hypothetical purchase task, participants will complete multiple trials where the price of a product will increase progressively. The availability of alternative products will be manipulated. We will measure demand elasticity (alpha) while product prices increase across trials.
Own-price and cross-price demand breakpoint | Day 1
  Participants will complete purchasing trials in a hypothetical purchase task. In the hypothetical purchase task, participants will complete multiple trials where the price of a product will increase progressively. The availability of alternative products will be manipulated. We will measure demand brekapoint while product prices increase across trials.
Own-price and cross-price demand Pmax | Day 1
  Participants will complete purchasing trials in a hypothetical purchase task. In the hypothetical purchase task, participants will complete multiple trials where the price of a product will increase progressively. The availability of alternative products will be manipulated. We will measure demand Pmax while product prices increase across trials.
Experimental Tobacco Marketplace purchase patterns | Day 1
  Participants will complete the Experimental Tobacco Marketplace (ETM) which is a virtual store designed to mimic real-world shopping environments. In the ETM participants will complete purchasing trials simulating different policy scenarios. We will measure quantity of products purchased per trial and number of individuals purchasing at least one product in each trial.

CONTACTS AND LOCATIONS:
Overall Officials: Roberta Freitas-Lemos, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

REFERENCES:
- [Background] Pickworth WB, Moolchan ET, Berlin I, Murty R. Sensory and physiologic effects of menthol and non-menthol cigarettes with differing nicotine delivery. Pharmacol Biochem Behav. 2002 Jan-Feb;71(1-2):55-61. doi: 10.1016/s0091-3057(01)00623-2. PMID 11812507
- [Background] Kyriakos CN, Driezen P, Fong GT, Chung-Hall J, Hyland A, Geboers C, Craig LV, Willemsen MC, Filippidis FT. Illicit purchasing and use of flavour accessories after the European Union menthol cigarette ban: findings from the 2020-21 ITC Netherlands Surveys. Eur J Public Health. 2023 Aug 1;33(4):619-626. doi: 10.1093/eurpub/ckad049. PMID 37527828
- [Background] Erinoso O, Clegg Smith K, Iacobelli M, Saraf S, Welding K, Cohen JE. Global review of tobacco product flavour policies. Tob Control. 2020 May 15;30(4):373-9. doi: 10.1136/tobaccocontrol-2019-055454. Online ahead of print. PMID 32414867
- [Background] Bandi P, Newton C, Xue Z, Thomson B, Asare S, Patel M, Islami F, Nargis N, Patel AV, Jemal A, Westmaas JL, Diver WR. Association of menthol-flavoured cigarette smoking with all-cause and cause-specific mortality risk. Tob Control. 2025 Feb 13:tc-2024-059020. doi: 10.1136/tc-2024-059020. Online ahead of print. PMID 39947700
- [Background] Lortet-Tieulent J, Goding Sauer A, Siegel RL, Miller KD, Islami F, Fedewa SA, Jacobs EJ, Jemal A. State-Level Cancer Mortality Attributable to Cigarette Smoking in the United States. JAMA Intern Med. 2016 Dec 1;176(12):1792-1798. doi: 10.1001/jamainternmed.2016.6530. PMID 27775761
- [Background] Havermans A, Pauwels CGGM, Bakker-'t Hart IME, Fayokun R, van Nierop LE, Hellmich IM, Talhout R. Across the world availability of flavour accessories for tobacco products. Tob Control. 2025 Jul 31;34(4):532-538. doi: 10.1136/tc-2023-058255. PMID 38580443